CLINICAL TRIAL: NCT02202590
Title: Pilot Study to Image the Esophagus Using Spectrally Encoded Confocal Microscopy (SECM)
Brief Title: Using Spectrally Encoded Confocal Microscopy (SECM) to Image the Esophagus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-P000863; 5R01DK091923-03 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-07-29 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: SECM; Esophagus; Eosinophilic Esophagitis; Allergy
MeSH Terms: conditions — Eosinophilic Esophagitis; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Imaging (Experimental): Participant will swallow the SECM capsule and Imaging will be performed using the SECM Imaging system.
  Interventions: Device: SECM Capsule

INTERVENTIONS:
Device: SECM Capsule — Imaging of the esophagus using the SECM capsule and system

SUMMARY:
The goal of this study is to test the feasibility and the tolerability of a tethered spectrally encoded confocal microscopy (SECM) capsule and to use it to image the esophagus.

DETAILED DESCRIPTION:
96 participants including healthy volunteers, patients with a suspicion of having Eosinophilic Esophagitis (EoE) and patients with a current or prior clinical diagnosis of EoE will be recruited and asked to swallow the SECM capsule while being awake and unsedated. The capsule is attached to a tether which allows the operator to control as well as navigate the capsule as it progresses down the esophagus using natural propulsive force called peristalsis.

As the capsule progresses, multiple 2-dimensional cross-sectional images of the esophagus are acquired. Images are analyzed at a later stage.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a healthy volunteer
* OR participant must have a suspicion of EoE
* OR participant must have a prior clinical suspicion of EoE
* Participant must be older than 14 years of age
* Participant must be able to give informed consent

Exclusion Criteria:

* Participants with the inability to swallow pills and capsules.
* Esophageal fistula and/or esophageal strictures with a stricture diameter that is smaller than the diameter of the capsule.
* Participants with prior endoscopic ablation or resection treatment of Barrett's Esophagus (BE)

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
SECM Imaging quality. Assessed qualitative values like resolution, tissue architecture, background scatter etc. | A single 20 minute visit (5-7 minute imaging).
  An investigator will qualitatively assess the the Feasibility of SECM Capsule and Imaging in EoE participant versus Healthy Controls. He will assess the quality of the recorded images and movies obtained with each exam after the imaging is completed. The images obtained by the SECM Capsule will be compared to the images obtained by clinical endoscopy if available.
Tolerability of SECM Capsule Imaging Procedure in Healthy and EoE Participant, measured by feedback scores. | Questionnaire adminstered directly after the imaging portion has been completed.
  After participating in the study, the participants will be asked for feedback about tolerability of the procedure using a questionnaire. This entails questions about discomfort levels and the participants ability to tolerate the tether and capsule during the whole and parts of the procedures. using a 0 -10 scale, participants will score how comfortable the procedure was during each stage. 10 being the most discomfort and 0 being the least discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No